CLINICAL TRIAL: NCT05945277
Title: Effectiveness of the Critical Time Intervention-Peer Support (CTI-PS) Model for Persons With Serious Mental Illness Discharged From Inpatient Psychiatric Treatment Facilities in Portugal
Brief Title: Critical Time Intervention-Peer Support
Acronym: CTI-PS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lisbon Institute of Global Mental Health - LIGMH (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTI-PS
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Psychotic Disorders; Schizophrenia; Bipolar Disorder; Schizo Affective Disorder
Keywords: Recovery; Peer support; Severe mental illness
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Critical Time Intervention - Peer Support

INTERVENTIONS:
Behavioral: Critical Time Intervention - Peer Support — CTI-PS is a time-limited, 9-month long intervention, provided at the critical time when a person is discharged from an inpatient psychiatric treatment facility.
  Arms: Intervention

SUMMARY:
There is increasing awareness of the importance of providing mental health services and support that promote a recovery-oriented and human rights-based approach. A mental health service system that is guided by a rehabilitation and recovery perspective places emphasis on treating the consequences of the illness rather than just the illness "per se", and on empowering people to regain control of their identity and life, and to have hope for the future. Within this philosophy, mental health policies in several countries advocate for the introduction of peer workers in mental health services, people with lived experience of mental health issues and recovery, who are employed to use their lived experience to support those who access mental health services. However, more effectiveness and implementation research is needed. Evidence also suggests that the period following hospital discharge is of high risk of treatment dropout for people with serious mental illness, thus interrupting their recovery process. Therefore, this vulnerable population may particularly benefit from more targeted interventions during this transitional period.

The research project will conduct a pilot randomized controlled trial to evaluate the feasibility, implementation and potential effectiveness of the Critical Time Intervention-Peer Support model, a recovery-oriented based model for people with serious mental illness discharged from inpatient psychiatric treatment facilities in Portugal. The randomized controlled trial (RCT) will be conducted in three psychiatric services in the Lisbon Metropolitan Area and their catchment areas. People with diagnoses of psychotic disorders discharged from inpatient psychiatric treatment facilities will be recruited and randomly divided into CTI-PS intervention or usual care. Those allocated to the intervention group will additionally receive CTI-PS rather than usual care alone over a 9-month period. Outcomes at baseline, 9- and 18-months will be analyzed by multilevel models, considering the observations clustered within sites. Longitudinal analyses will be used to examine trends over time of the outcomes of interest.

The implementation of the CTI-PS model will introduce a novel approach to community mental health care that has not yet been tried in Portugal. This study aims to explore to what extent this intervention can be effectively implemented in countries with the characteristics of Portugal. Additionally, the proposed research aims to contribute to the global knowledge about peer interventions by exploring whether the CTI model can maintain its effectiveness using peers.

DETAILED DESCRIPTION:
Critical Time Intervention-Peer Support is delivered by Community Mental Health Workers (CMHWs) and Peer Support Workers (PSWs). They will be selected, recruited, and trained by members of the research team to deliver mental health care according to the manualized recovery-oriented program. Ongoing regular supervision of PSWs and CMHWs, in weekly meetings, will be conducted throughout the study by members of the research team trained in CTI-PS by those who originally developed it at the Columbia University.

Those allocated to the intervention group will receive usual care and, in addition, CTI-PS services over a 9-month period.

The intervention has two broad objectives: 1) to collaborate with participants to develop durable connections to support systems, including both formal and informal supports (e.g., mental health services, primary care clinics, family, and friends); and 2) to provide practical and emotional support, helping the individual to overcome a critical period of transition during which they can feel especially vulnerable.

The work of CTI-PS will focus on areas identified as crucial for strengthening the individual's continuum of services and forming enduring links with their community supports. The phases of CTI are Initiation, Try-Out, and Transfer of Care. The PSW-CMHW will collaborate with the participants to identify barriers to their recovery and develop a sustainable plan to engage in and use community supports and resources during and after CTI. They will also use their knowledge to increase participants' autonomy, strengthen their connection to health services, and expand their support networks. The role of CTI workers is specifically designed to avoid becoming the primary source of care for the individual.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* Any psychotic disorder diagnosis based on the International Classification of Diseases - 10th revision (ICD-10) criteria, including both non-affective (e.g., schizophrenia) and affective psychosis (e.g., bipolar disorder)
* Having been discharged from inpatient psychiatric treatment facilities in the month prior to recruitment

Exclusion Criteria:

* Active suicidal ideation.
* Cognitive, neurological, or other sensorial conditions likely to preclude or affect an objective assessment via interview procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
WHOQOL-BREF | 18 months
  Health-related quality of life, assessed by the WHO Quality of Life Scale - Brief Version (WHOQOL-BREF). This instrument has 26 items and measures the following domains: physical and psychological health, social relationships, and environment, with two additional general questions.
Camberwell Assessment of Need (CAN) | 18 months
  Unmet needs, assessed by the Camberwell Assessment of Need (CAN), which evaluates 22 areas of need such as accommodation, food, safety to self, among others.

SECONDARY OUTCOMES:
Psychopathology, assessed by the Brief Psychiatric Rating Scale (BPRS) | 18 months
Level of disability, assessed by the WHO Disability Assessment Schedule (WHODAS 2.0) | 18 months
Orientation toward recovery, assessed by the INSPIRE - Research Into Recovery | 18 months
Self-stigma, assessed by the Internalized Stigma of Mental Illness (ISMI) | 18 months
Substance use, assessed by the WHO Alcohol, Smoking and Substance Involvement Screening Test Schedule (WHO ASSIST) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Silva, M.D., PhD, Principal Investigator — Lisbon Institute of Global Mental Health
Locations (3):
- Portugal (3):
  - Centro Hospitalar Lisboa Ocidental, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, Lisbon
  - Hospital Beatriz Ângelo, Loures

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.criticaltime.org/cti-model/
- See also: Related Info — http://lisboninstitutegmh.org